CLINICAL TRIAL: NCT00666406
Title: Pharmacokinetic Comparison of Advate rAHF-PFM With Recombinate rAHF in Patients With Severe Hemophilia A: a Phase IV, Prospective, Randomized, Controlled, Cross-over, Single Center Study
Brief Title: Pharmacokinetic Comparison of Advate rAHF-PFM With Recombinate rAHF in Patients With Severe Hemophilia A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 060601; 2007-004834-18 (EudraCT Number)
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Results first posted 2013-03-26 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Advate rAHF-PFM
  Interventions: Drug: Antihemophilic Factor (Recombinant) - Plasma/Albumin Free Method (rAHF-PFM)
- 2 (Active Comparator): Recombinate rAHF
  Interventions: Drug: Recombinant Factor VIII (rAHF)

INTERVENTIONS:
Drug: Antihemophilic Factor (Recombinant) - Plasma/Albumin Free Method (rAHF-PFM) — Infusion of 50 +/- 5 IU/kg bodyweight
  Other Names: Advate rAHF-PFM; Recombinant Protein-Free Factor VIII (rAHF-PFM)
  Arms: 1
Drug: Recombinant Factor VIII (rAHF) — Infusion of 50 +/- 5 IU/kg bodyweight
  Other Names: Recombinate rAHF; Antihemophilic Factor (Recombinant)
  Arms: 2

SUMMARY:
The purpose of this study is to compare the pharmacokinetic parameters and safety of Advate rAHF-PFM versus Recombinate rAHF in well described previously treated patients with severe hemophilia A (factor VIII level < 1%).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained from participant or legally authorized representative
* 15-60 years old
* Factor VIII level < 1% as documented by previously measured factor VIII and genotyping
* Previously treated with factor VIII concentrate(s) for a minimum of at least 150 exposure days (as documented by the study site investigator) prior to study entry
* Observed decrease of efficacy by subject and/or treating physician after being switched from Recombinate rAHF to Advate rAHF-PFM

Exclusion Criteria:

* The participant has a detectable factor VIII inhibitor at screening, with a titer >= 0.4 Bethesda Unit (BU) (Nijmegen modification of the Bethesda Assay) measured at the local and the central laboratory
* The participant has a known hypersensitivity to mouse or hamster proteins
* The participant is participating in another investigational drug study within 30 days prior to screening
* The participant is identified by the investigator as being unable or unwilling to cooperate with study procedures

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2008-03-31 (Actual); Primary Completion 2009-02-18 (Actual); Study Completion 2009-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Bonn, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 unique participants enrolled and treated at a single study site in Germany
Pre-assignment Details: Participants required a factor VIII (FVIII) washout period ≥48 hours before receiving any pharmacokinetic (PK) infusions and could not be actively bleeding at the time of the infusion.
Groups:
- Advate rAHF-PFM Then Recombinate rAHF: First infusion - Advate Antihemophilic Factor (Recombinant)-Plasma/Albumin Free Method (rAHF-PFM): Infusion of 50 +/- 5 IU/kg bodyweight Second infusion - Recombinate Antihemophilic Factor (Recombinant) (rAHF): Infusion of 50 +/- 5 IU/kg bodyweight
- Recombinate rAHF Then Advate rAHF-PFM: First infusion - Recombinate rAHF: Infusion of 50 +/- 5 IU/kg bodyweight Second infusion - Advate rAHF-PFM: Infusion of 50 +/- 5 IU/kg bodyweight
Period: First PK Infusion
Arm/Group | Advate rAHF-PFM Then Recombinate rAHF | Recombinate rAHF Then Advate rAHF-PFM
Started | 6 | 3
Completed | 6 | 3
Not Completed | 0 | 0
Period: Second PK Infusion
Arm/Group | Advate rAHF-PFM Then Recombinate rAHF | Recombinate rAHF Then Advate rAHF-PFM
Started | 6 | 3
Completed | 6 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes groups randomized to receive Advate rAHF-PFM and Recombinate rAHF first.
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 9

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From 0 to 48 Hours. One-Stage Activated Partial Thromboplastin Time (aPTT) -Based Assay Performed at Central Laboratory (Medical University Vienna)
Description: AUC estimated by linear trapezoidal method. The linear trapezoidal method is a numerical method used to approximate the area under a curve.
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: IU*h/dL
Groups:
- Advate rAHF-PFM: Advate rAHF-PFM: Infusion of 50 +/- 5 IU/kg bodyweight
- Recombinate rAHF: Recombinate rAHF: Infusion of 50 +/- 5 IU/kg bodyweight
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
IU*h/dL | 1104 [950 to 1328] | 1294 [1149 to 1536]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.173, 90% CI 2-sided [1.089 to 1.262]

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From 0 to 48 Hours. Chromogenic Assay Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: as for outcome 1
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: IU*h/dL
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
IU*h/dL | 1180 [999 to 1497] | 1358 [1146 to 1547]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.139, 90% CI 2-sided [1.043 to 1.243]

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From 0 to 48 Hours. FVIII One-Stage Clotting Assay (Bonn Method) Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: as for outcome 1
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: IU*h/dL
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
IU*h/dL | 833 [697 to 970] | 901 [629 to 1070]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.060, 90% CI 2-sided [0.866 to 1.297]

4. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From 0 to 48 Hours. FVIII Clotting Assay. Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: as for outcome 1
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: IU*h/dL
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
IU*h/dL | 1505 [1215 to 1741] | 1664 [1340 to 1911]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.071, 90% CI 2-sided [0.972 to 1.179]

5. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From 0 to Infinity. One-Stage aPTT-Based Assay Performed at Central Laboratory (Medical University Vienna)
Description: AUC estimated by linear trapezoidal method. The linear trapezoidal method is a numerical method used to approximate the area under a curve. FVIII activity measurement
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: IU*h/dL
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
IU*h/dL | 1190 [1031 to 1360] | 1393 [1232 to 1574]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.171, 90% CI 2-sided [1.099 to 1.247]

6. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From 0 to Infinity. Chromogenic Assay Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: as for outcome 1
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: IU*h/dL
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
IU*h/dL | 1282 [1037 to 1626] | 1452 [1137 to 1696]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.135, 90% CI 2-sided [1.092 to 1.180]

7. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From 0 to Infinity. FVIII One-Stage Clotting Assay (Bonn Method) Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: as for outcome 1
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: IU*h/dL
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
IU*h/dL | 874 [734 to 1031] | 926 [655 to 1152]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.036, 90% CI 2-sided [0.857 to 1.253]

8. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From 0 to Infinity. FVIII Clotting Assay. Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: as for outcome 1
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: IU*h/dL
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
IU*h/dL | 1598 [1340 to 1923] | 1731 [1453 to 2162]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.093, 90% CI 2-sided [1.007 to 1.186]

9. Secondary Outcome: Systemic Clearance (Cl). One-Stage aPTT-Based Assay Performed at Central Laboratory (Medical University Vienna)
Description: Systemic clearance in mL/kg/h will be calculated as the dose in IU/kg divided by the total area under the curve.
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: mL/h/kg
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
mL/h/kg | 4.31 [3.92 to 4.85] | 3.68 [3.41 to 4.19]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 0.854, 90% CI 2-sided [0.798 to 0.913]

10. Secondary Outcome: Systemic Clearance (Cl). Chromogenic Assay Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: Systemic clearance in mL/kg/h will be calculated as the dose in IU/kg divided by the total area under the curve.
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: mL/h/kg
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
mL/h/kg | 4.00 [3.28 to 4.88] | 3.53 [3.03 to 4.43]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 0.881, 90% CI 2-sided [0.847 to 0.916]

11. Secondary Outcome: Systemic Clearance (Cl). FVIII One-Stage Clotting Assay (Bonn Method) Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: Systemic clearance in mL/kg/h will be calculated as the dose in IU/kg divided by the total area under the curve.
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: mL/h/kg
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
mL/h/kg | 5.87 [4.40 to 7.35] | 5.53 [4.28 to 8.19]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 0.964, 90% CI 2-sided [0.799 to 1.164]

12. Secondary Outcome: Systemic Clearance (Cl). FVIII Clotting Assay. Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: Systemic clearance in mL/kg/h will be calculated as the dose in IU/kg divided by the total area under the curve.
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: mL/h/kg
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
mL/h/kg | 3.21 [2.63 to 3.85] | 2.96 [2.35 to 3.79]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 0.915, 90% CI 2-sided [0.841 to 0.995]

13. Secondary Outcome: Maximum Plasma Concentration (C-max). One-Stage aPTT-Based Assay Performed at Central Laboratory (Medical University Vienna)
Description: C-max will be calculated as the maximum concentration following infusion of either Advate or Recombinate.
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: IU/dL
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
IU/dL | 93 [74 to 112] | 108 [91 to 130]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.177, 90% CI 2-sided [1.104 to 1.256]

14. Secondary Outcome: Maximum Plasma Concentration (C-max). Chromogenic Assay Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: C-max will be calculated as the maximum concentration following infusion of either Advate or Recombinate.
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: IU/dL
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
IU/dL | 104 [79 to 148] | 119 [104 to 144]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.152, 90% CI 2-sided [1.039 to 1.277]

15. Secondary Outcome: Maximum Plasma Concentration (C-max). FVIII One-Stage Clotting Assay (Bonn Method) Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: C-max will be calculated as the maximum concentration following infusion of either Advate or Recombinate.
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: IU/dL
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
IU/dL | 78 [66 to 100] | 94 [72 to 149]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.182, 90% CI 2-sided [1.029 to 1.359]

16. Secondary Outcome: Maximum Plasma Concentration (C-max). FVIII Clotting Assay. Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: C-max will be calculated as the maximum concentration following infusion of either Advate or Recombinate.
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: IU/dL
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
IU/dL | 100 [72 to 121] | 112 [92 to 137]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.133, 90% CI 2-sided [1.010 to 1.270]

17. Secondary Outcome: Terminal Half-life. One-Stage aPTT-Based Assay Performed at Central Laboratory (Medical University Vienna)
Description: Computed from the terminal or disposition rate constant obtained from log-linear fitting using the least squares deviation to the last five quantifiable concentrations (9 to 48 hours).
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: hours
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
hours | 10.7 [8.3 to 12.8] | 10.9 [9.1 to 13.1]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.008, 90% CI 2-sided [0.969 to 1.050]

18. Secondary Outcome: Terminal Half-life. Chromogenic Assay Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: Computed from the terminal or disposition rate constant obtained from log-linear fitting using the least squares deviation to the last five quantifiable concentrations.
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: hours
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
hours | 11.7 [8.5 to 13.5] | 10.8 [8.2 to 12.2]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 0.964, 90% CI 2-sided [0.843 to 1.102]

19. Secondary Outcome: Terminal Half-life. FVIII One-Stage Clotting Assay (Bonn Method) Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: as for outcome 18
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: hours
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
hours | 9.5 [7.5 to 12.8] | 9.9 [7.6 to 11.5]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.038, 90% CI 2-sided [0.926 to 1.163]

20. Secondary Outcome: Terminal Half-life. FVIII Clotting Assay. Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: as for outcome 18
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: hours
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
hours | 12.4 [9.3 to 14.2] | 12.1 [8.9 to 13.9]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.015, 90% CI 2-sided [0.901 to 1.144]

21. Secondary Outcome: Incremental Recovery. One-Stage aPTT-Based Assay Performed at Central Laboratory (Medical University Vienna)
Description: Increase in factor VIII concentration from pre- to post-infusion.
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: (IU/dL)/(IU/kg)
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
(IU/dL)/(IU/kg) | 1.81 [1.52 to 2.10] | 2.11 [1.89 to 2.42]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.178, 90% CI 2-sided [1.106 to 1.254]

22. Secondary Outcome: Incremental Recovery. Chromogenic Assay Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: Computed from the terminal or disposition rate constant obtained from log_e -linear fitting using the least squares deviation to the last five quantifiable concentrations.
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: (IU/dL)/(IU/kg)
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
(IU/dL)/(IU/kg) | 2.04 [1.53 to 2.70] | 2.33 [2.02 to 2.69]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.152, 90% CI 2-sided [1.038 to 1.279]

23. Secondary Outcome: Incremental Recovery. FVIII One-Stage Clotting Assay (Bonn Method) Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: Increase in factor VIII concentration from pre- to post-infusion
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: (IU/dL)/(IU/kg)
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
(IU/dL)/(IU/kg) | 1.53 [1.24 to 1.82] | 1.84 [1.49 to 2.82]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.183, 90% CI 2-sided [1.027 to 1.362]

24. Secondary Outcome: Incremental Recovery. FVIII Clotting Assay. Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: Increase in factor VIII concentration from pre- to post-infusion
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: (IU/dL)/(IU/kg)
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
(IU/dL)/(IU/kg) | 1.94 [1.44 to 2.27] | 2.19 [1.74 to 2.64]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.133, 90% CI 2-sided [1.012 to 1.270]

25. Secondary Outcome: Mean Residence Time (MRT). One-Stage aPTT-Based Assay Performed at Central Laboratory (Medical University Vienna)
Description: The MRT in hours will be calculated as total area under the moment curve divided by the total area under the curve.
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: Hours
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
Hours | 14.1 [11.0 to 17.5] | 14.4 [12.1 to 17.6]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.009, 90% CI 2-sided [0.964 to 1.056]

26. Secondary Outcome: Mean Residence Time (MRT). Chromogenic Assay Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: The MRT in hours will be calculated as total area under the moment curve divided by the total area under the curve.
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: Hours
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
Hours | 15.1 [10.9 to 18.6] | 14.2 [10.3 to 16.2]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 0.971, 90% CI 2-sided [0.849 to 1.112]

27. Secondary Outcome: Mean Residence Time (MRT). FVIII One-Stage Clotting Assay (Bonn Method) Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: The MRT in hours will be calculated as total area under the moment curve divided by the total area under the curve.
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: Hours
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
Hours | 12.5 [9.1 to 16.7] | 12.8 [10.1 to 16.4]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.020, 90% CI 2-sided [0.938 to 1.109]

28. Secondary Outcome: Mean Residence Time (MRT). FVIII Clotting Assay. Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: The MRT in hours will be calculated as total area under the moment curve divided by the total area under the curve.
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: Hours
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
Hours | 17.3 [12.4 to 19.6] | 16.9 [13.2 to 19.6]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 0.996, 90% CI 2-sided [0.894 to 1.111]

29. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax). One-Stage aPTT-Based Assay Performed at Central Laboratory (Medical University Vienna)
Description: Tmax in hours was defined as the minimum time to reach Maximum plasma concentration (Cmax).
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: Hours
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
Hours | 0.25 [0.25 to 0.25] | 0.25 [0.25 to 0.25]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.000, 90% CI 2-sided [1.000 to 1.000]

30. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax). Chromogenic Assay Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: Tmax in hours was defined as the minimum time to reach Maximum plasma concentration (Cmax).
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: Hours
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
Hours | 0.31 [0.25 to 0.50] | 0.42 [0.25 to 1.00]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.303, 90% CI 2-sided [0.841 to 2.020]

31. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax). FVIII One-Stage Clotting Assay (Bonn Method) Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: Tmax in hours was defined as the minimum time to reach Maximum plasma concentration (Cmax).
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: Hours
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
Hours | 0.45 [0.25 to 1.00] | 0.31 [0.25 to 0.50]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 0.724, 90% CI 2-sided [0.304 to 1.728]

32. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax). FVIII Clotting Assay. Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: Tmax in hours was defined as the minimum time to reach Maximum plasma concentration (Cmax).
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: Hours
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
Hours | 0.38 [0.25 to 1.00] | 0.51 [0.25 to 3.00]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 1.059, 90% CI 2-sided [0.442 to 2.539]

33. Secondary Outcome: Volume of Distribution at Steady State (Vss). One-Stage aPTT-Based Assay Performed at Central Laboratory (Medical University Vienna)
Description: Computed as weight-adjusted Clearance * Mean Residence Time
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: mL/kg
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
mL/kg | 60.8 [48.2 to 75.7] | 52.9 [43.9 to 62.0]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 0.862, 90% CI 2-sided [0.807 to 0.920]

34. Secondary Outcome: Volume of Distribution at Steady State (Vss). Chromogenic Assay Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: Computed as weight-adjusted Clearance (CL) * Mean Residence Time
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: mL/kg
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
mL/kg | 60.4 [45.5 to 76.6] | 50.2 [45.4 to 58.2]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 0.855, 90% CI 2-sided [0.730 to 1.002]

35. Secondary Outcome: Volume of Distribution at Steady State (Vss). FVIII One-Stage Clotting Assay (Bonn Method) Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: Computed as weight-adjusted CL * Mean Residence Time
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: mL/kg
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
mL/kg | 73.2 [54.6 to 87.5] | 70.9 [67.5 to 89.5]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 0.984, 90% CI 2-sided [0.788 to 1.228]

36. Secondary Outcome: Volume of Distribution at Steady State (Vss). FVIII Clotting Assay. Performed at Local Laboratory (i.e., University of Bonn, the Study Site)
Description: Computed as weight-adjusted CL * Mean Residence Time
Time Frame: 0-30 minutes before infusion up to 48 hours post-infusion
Population: All enrolled participants
Measure: Geometric Mean (90% Confidence Interval); unit: mL/kg
Arm/Group | Advate rAHF-PFM | Recombinate rAHF
Number analyzed (Participants) | 9 | 9
mL/kg | 55.6 [40.4 to 69.1] | 50.0 [39.8 to 63.8]
Statistical Analysis 1: Comparison: Advate rAHF-PFM vs Recombinate rAHF; Test type: Superiority or Other; Ratio of the geometric means = 0.911, 90% CI 2-sided [0.800 to 1.039]

ADVERSE EVENTS:
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter requires a review of results communications (e.g., for confidential information and/or manuscript amendment proposals which do not negatively influence the scientific character of impartiality) ≥30 days prior to submission or communication. Baxter may request an additional delay of ≤60 days (e.g., for intellectual property protection)